CLINICAL TRIAL: NCT03698019
Title: A Phase II Randomized Study of Adjuvant Versus NeoAdjuvant Pembrolizumab (MK-3475) for Clinically Detectable Stage III-IV High-Risk Melanoma
Brief Title: A Study to Compare the Administration of Pembrolizumab After Surgery Versus Administration Both Before and After Surgery for High-Risk Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-02107; NCI-2018-02107 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1801 (Other: SWOG); S1801 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Acral Lentiginous Melanoma; Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Mucosal Melanoma
MeSH Terms: interventions — Specimen Handling; Magnetic Resonance Spectroscopy; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (adjuvant pembrolizumab) (Experimental): Within 17 days (preferably within 14 days) days after IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 18 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood throughout the study and MRI or CT on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Procedure: Therapeutic Conventional Surgery
- Arm II (adjuvant and neoadjuvant pembrolizumab) (Active Comparator): Patients receive pembrolizumab IV over 30 minutes on day 1 every 3 weeks for 3 cycles, then undergo surgery within 3 weeks. Within 84 days, patients receive pembrolizumab IV over 30 minutes every 3 weeks for 15 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood throughout the study and MRI or CT on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This phase II trial studies how pembrolizumab works before and after surgery in treating patients with stage III-IV high-risk melanoma. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving pembrolizumab before and after surgery may work better compared to after surgery alone in treating melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare event-free survival (EFS) in participants with high-risk resectable melanoma randomized to neoadjuvant pembrolizumab (MK-3475) with participants randomized to adjuvant pembrolizumab (MK-3475).

SECONDARY OBJECTIVES:

I. To assess the frequency and severity of toxicities on each of the arms. II. To compare between arms overall survival (OS), disease control at 24 weeks, locoregional control in the surgical site(s), and total number of pembrolizumab (MK-3475) doses received.

III. On the neoadjuvant arm, to estimate the pathologic response rate, the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 response rate (confirmed and unconfirmed complete response [CR] and partial response [PR]), and the immune-related (i)RECIST response rate (confirmed and unconfirmed CR and PR), before surgical resection; to compare definitions of pathologic partial response; and to evaluate the association between pathologic response and EFS and OS.

IV. To describe the proportion of participants on each arm who received the surgery planned at randomization.

ADDITIONAL OBJECTIVE:

I. To bank tumor tissue and whole blood in anticipation of future correlative studies in this participant population.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Within 17 days (preferably within 14 days) days after surgical resection, patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 3 weeks for 18 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood throughout the study, and magnetic resonance imaging (MRI) or computers tomography (CT) on study.

ARM II: Patients receive pembrolizumab IV over 30 minutes on day 1 every 3 weeks for 3 cycles, then undergo surgical resection within 3 weeks. Within 84 days, patients receive pembrolizumab IV over 30 minutes every 3 weeks for 15 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood throughout the study and MRI or CT on study.

After completion of study treatment, patients are followed up at 3 and 12 weeks, then every 3 months for 2 years, every 6 months for 3 years, then every 12 months for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1 REGISTRATION (RANDOMIZATION): Patients must have clinically detectable stage III (clinically detectable N1b, N1c, N2b, N2c, N3b and N3c) or stage IV resectable melanoma. Patients with melanoma of mucosal or acral origin are eligible. Patients with melanoma of uveal origin are not eligible. Patients with a history of brain metastases are not eligible. Clinically detectable is defined as disease that is apparent and measurable via physical examination or radiographic imaging.
* STEP 1 REGISTRATION (RANDOMIZATION): Patients are eligible for this trial either at initial presentation of their melanoma or at the time of the first detected nodal, satellite/in-transit, distant metastases, or recurrent disease in prior lymphadenectomy basin or distant site. Nodal, satellite/in-transit metastasis, distant metastases or disease in a prior complete lymphadenectomy basin must have been confirmed histologically by hematoxylin (H) & eosin (E) stained slides.
* STEP 1 REGISTRATION (RANDOMIZATION): Patients with multiple regional nodal basin involvement are eligible. Gross or microscopic extracapsular nodal extension is permitted.
* STEP 1 REGISTRATION (RANDOMIZATION): Patients must have histologically proven stage IIIB or higher. This would entail pathologic confirmation beyond the primary or initial diagnosis of melanoma involving fine needle aspiration cytology or biopsy confirmation of any N-category or M-category resectable site.
* STEP 1 REGISTRATION (RANDOMIZATION): Patients must not have received previous neoadjuvant treatment for their melanoma. Patients may have received prior non-immunotherapy adjuvant therapy. Patients must not have had prior immunotherapy including, but not limited to ipilimumab, interferon alfa-2b, high dose interleukin (IL)-2, pegylated-interferon (PEG-IFN), anti-PD-1, anti-PD-L1 intra-tumoral, or vaccine therapies. Patients must not be planning to receive any of the prohibited therapies during treatment phases on the study.
* STEP 1 REGISTRATION (RANDOMIZATION): Patients must not be planning to receive concomitant other biologic therapy, hormonal therapy, other chemotherapy, surgery, while on protocol therapy.
* STEP 1 REGISTRATION (RANDOMIZATION): Patients may have received prior radiation therapy, including after prior surgical resection. All adverse events associated with prior surgery and radiation therapy must have resolved to =< grade 1 prior to randomization.
* STEP 1 REGISTRATION (RANDOMIZATION): Patients must be >= 18 years of age
* STEP 1 REGISTRATION (RANDOMIZATION): All patients must have disease status documented by a complete physical examination and imaging studies within 42 days prior to randomization. Imaging studies must include a CT of the chest, abdomen and pelvis with intravenous contrast (unless contraindicated). For patients with melanoma arising from the head and neck, dedicated neck imaging (CT with intravenous contrast is required. If the patient has unknown primary with disease in the axilla, neck imaging is required CT imaging must be done with intravenous contrast if there are no contraindications for it. Extremity melanomas must be imaged using CT with intravenous contrast or MRI with and without gadolinium

  * Note: PET-CT scans are NOT acceptable to establish eligibility. Non-iodinated CT scans that are part of common PET-CT imaging protocols do not provide contrast for difficult to ascertain areas such as the neck and liver, and do not provide enough CT detail to perform appropriate RECIST 1.1 measurements. As such, a PET-CT with non-contrast CT or non-diagnostic quality CT images is considered insufficient for the detection of melanoma.
* STEP 1 REGISTRATION (RANDOMIZATION): All patients must have a CT or magnetic resonance imaging (MRI) of the brain within 42 days prior to randomization. The brain CT or MRI should be performed with intravenous contrast (unless contraindicated).
* STEP 1 REGISTRATION (RANDOMIZATION): Absolute neutrophil count (ANC) >= 1,500/microliter (mcL) (within 42 days prior to randomization).
* STEP 1 REGISTRATION (RANDOMIZATION): Platelets >= 100,000/mcL (within 42 days prior to randomization).
* STEP 1 REGISTRATION (RANDOMIZATION): Hemoglobin >= 10 g/dL (within 42 days prior to randomization).
* STEP 1 REGISTRATION (RANDOMIZATION): Total bilirubin =< 1.5 x institutional upper limit of normal (IULN) (except patients with Gilbert's syndrome, who must have a total bilirubin < 3.0 mg/dL) (within 42 days prior to randomization).
* STEP 1 REGISTRATION (RANDOMIZATION): Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2 x IULN (within 42 days prior to randomization).
* STEP 1 REGISTRATION (RANDOMIZATION): Alkaline phosphatase =< 2 x IULN (within 42 days prior to randomization).
* STEP 1 REGISTRATION (RANDOMIZATION): Patients must have lactate dehydrogenase (LDH) performed within 42 days prior to randomization.
* STEP 1 REGISTRATION (RANDOMIZATION): Patients must have adequate renal function as evidenced by calculated creatinine clearance > 30 mL/min. The creatinine level (mg/dL) used in the calculation must be obtained within 42 days prior to randomization.
* STEP 1 REGISTRATION (RANDOMIZATION): Patients must have Zubrod performance status =< 2.
* STEP 1 REGISTRATION (RANDOMIZATION): Patients must not have a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* STEP 1 REGISTRATION (RANDOMIZATION): Patients must not have an active infection requiring systemic therapy.
* STEP 1 REGISTRATION (RANDOMIZATION): Patients must not have active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* STEP 1 REGISTRATION (RANDOMIZATION): Patients must not have received live vaccines within 42 days prior to randomization. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, shingles, yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid (oral) vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed.

  * NOTE: The COVID-19 vaccines (currently available and those in the pipeline for FDA emergency use authorization or FDA approval) do not contain live virus, and therefore, COVID-19 vaccination does not affect or preclude eligibility for the S1801 trial. For patients who have undergone lymphadenectomy, vaccines should be delivered to a limb with an intact lymph node basin (Sentinel lymph node biopsy in a limb is acceptable). The vaccine should not be administered in a limb that has undergone lymphadenectomy.
* STEP 1 REGISTRATION (RANDOMIZATION): Patients known to be human immunodeficiency virus (HIV) positive are eligible if they meet the following criteria within 30 days prior to randomization: stable and adequate CD4 counts (>= 350 mm^3), and serum HIV viral load of < 25,000 IU/ml. Patients may be on or off anti-viral therapy so long as they meet the CD4 count criteria.
* STEP 1 REGISTRATION (RANDOMIZATION): Patients must not have known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection prior to randomization. Note: No testing for hepatitis B and hepatitis C is required unless mandated by local health authority.
* STEP 1 REGISTRATION (RANDOMIZATION): Prior malignancy is allowed providing it does not require concurrent therapy.
* STEP 1 REGISTRATION (RANDOMIZATION): Women of childbearing potential must have a negative urine or serum pregnancy test within 28 days prior to randomization. Women/men of reproductive potential must have agreed to use an effective contraceptive method for the course of the study through 120 days after the last dose of study medication. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. A woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy, or bilateral tubal ligation. However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures. Patients must not be pregnant or nursing due to unknown teratogenic side effects.
* STEP 1 REGISTRATION (RANDOMIZATION): Patients must be deemed medically fit to undergo surgery by the treating medical/surgical team.
* STEP 1 REGISTRATION (RANDOMIZATION): Patients must be willing to submit the following surgical specimens: either all tissue blocks from the surgical specimen or two slides per block ([1] hematoxylin and eosin [H&E] slide and [1] unstained slide OR [2] unstained slides if H&E stained slides cannot be provided).
* STEP 1 REGISTRATION (RANDOMIZATION): Patients must be offered the opportunity to participate in specimen banking.
* STEP 1 REGISTRATION (RANDOMIZATION): Patients must be informed of the investigational nature of this study and must sign and give written informed consent for this protocol in accordance with institutional and federal guidelines.
* STEP 1 REGISTRATION (RANDOMIZATION): As a part of the Oncology Patient Enrollment Network (OPEN) randomization process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system.
* STEP 2 REGISTRATION (SURGERY): Patients randomized to arm 2 (neoadjuvant arm) must be willing to submit tissue to determine pathologic response regardless of number of pre-operative doses of pembrolizumab (MK-3475) received. Determination of pathologic response cannot be done on less than the full surgical specimen.
* STEP 2 REGISTRATION (SURGERY): Patients must have disease assessments by CT chest/abdomen/pelvis with IV contrast, and neck CT with IV contrast if primary head and neck melanoma, performed within 42 days (and no more than 49 days) before the planned date of surgery. MRI combined with non-contrast CT is an acceptable alternative for patients with CT contrast allergy, but imaging must encompass total body.
* STEP 2 REGISTRATION (SURGERY): Patients must register to step 2 within 17 days prior to planned date of surgery.
* STEP 3 REGISTRATION (ADJUVANT THERAPY): Patients must have undergone surgery prior to Step 3 registration. The Step 2 surgery must have completely resected their melanoma.

  * Patients with gross positive residual disease following surgery do not qualify as having disease-free status, and, therefore, such patients are not eligible to register for adjuvant therapy.
  * Patients with microscopic residual disease (i.e., positive margins) can be treated with re-excision or radiation, per site discretion, to render the patient disease-free prior to registration of adjuvant therapy.
  * Disease-free status must be documented by a complete physical examination and radiographic imaging studies within 42 days prior to Step 3 registration. Imaging studies must include a CT of the chest, abdomen, and pelvis (unless contraindicated). Extremity melanomas must be imaged using CT with intravenous contrast or MRI with and without gadolinium. CT imaging must be done with intravenous contrast if there are no contraindications for it.
  * For patients with melanoma arising from the head and neck, dedicated neck imaging (CT with IV contrast, unless contraindicated) is required.
  * If the patient has had unknown primary with disease in the axilla, neck imaging is required to assure the region is clear of cancer.
  * Any other clinically indicated imaging studies if performed (e.g., bone scan) must show no evidence of disease.
* STEP 3 REGISTRATION (ADJUVANT THERAPY): Patients must be registered to step 3 no more than 84 days after date of surgery.
* STEP 3 REGISTRATION (ADJUVANT THERAPY): Patients with R0 or R1 resections must have disease-free status documented by a complete physical examination and imaging studies within 42 days prior to step 3 registration. These patients must have disease assessments by CT chest/abdomen/pelvis with IV contrast, and neck CT with IV contrast if primary head and neck melanoma. MRI combined with non-contrast CT is an acceptable alternative for patients with CT contrast allergy, but imaging must encompass total body.
* STEP 3 REGISTRATION (ADJUVANT THERAPY): Patients with R2 resections are not eligible for step 3 and must be removed from study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2026-10-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sapna P Patel, Principal Investigator — SWOG Cancer Research Network
Locations (818):
- United States (818):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Banner Boswell Medical Center, Sun City, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Kaiser Permanente Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Keck Medicine of USC Huntington Beach, Huntington Beach, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Loma Linda Healthcare System, Loma Linda, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Providence Queen of The Valley, Napa, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Sutter Cancer Research Consortium, Novato, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Lutheran Hospital - Cancer Centers of Colorado, Golden, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - MercyOne Genesis Silvis Cancer Center, Silvis, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Franciscan Saint Elizabeth Health - Lafayette East, Lafayette, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Reid Health, Richmond, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - MercyOne Genesis Davenport Medical Center, Davenport, Iowa
  - MercyOne Genesis Davenport Cancer Center, Davenport, Iowa
  - Iowa Cancer Specialists, Davenport, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Our Lady of The Lake, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Ochsner Hematology Oncology North Shore - Covington (West Region), Covington, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Garnet Health Medical Center, Middletown, New York
  - University of Rochester, Rochester, New York
  - Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Wake Forest Baptist Health - Hematology Oncology - Statesville, Statesville, North Carolina
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Mount Carmel New Albany Surgical Hospital, New Albany, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Mercy Health Sylvania Radiation Oncology Center, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Portland VA Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Hendrick Medical Center, Abilene, Texas
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Franklin, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Ascension Saint Francis Hospital, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Long GV, Menzies AM, Scolyer RA. Neoadjuvant Checkpoint Immunotherapy and Melanoma: The Time Is Now. J Clin Oncol. 2023 Jun 10;41(17):3236-3248. doi: 10.1200/JCO.22.02575. Epub 2023 Apr 27. PMID 37104746
- [Derived] Patel SP, Othus M, Chen Y, Wright GP Jr, Yost KJ, Hyngstrom JR, Hu-Lieskovan S, Lao CD, Fecher LA, Truong TG, Eisenstein JL, Chandra S, Sosman JA, Kendra KL, Wu RC, Devoe CE, Deutsch GB, Hegde A, Khalil M, Mangla A, Reese AM, Ross MI, Poklepovic AS, Phan GQ, Onitilo AA, Yasar DG, Powers BC, Doolittle GC, In GK, Kokot N, Gibney GT, Atkins MB, Shaheen M, Warneke JA, Ikeguchi A, Najera JE, Chmielowski B, Crompton JG, Floyd JD, Hsueh E, Margolin KA, Chow WA, Grossmann KF, Dietrich E, Prieto VG, Lowe MC, Buchbinder EI, Kirkwood JM, Korde L, Moon J, Sharon E, Sondak VK, Ribas A. Neoadjuvant-Adjuvant or Adjuvant-Only Pembrolizumab in Advanced Melanoma. N Engl J Med. 2023 Mar 2;388(9):813-823. doi: 10.1056/NEJMoa2211437. PMID 36856617
- [Derived] Gorry C, McCullagh L, O'Donnell H, Barrett S, Schmitz S, Barry M, Curtin K, Beausang E, Barry R, Coyne I. Neoadjuvant treatment for stage III and IV cutaneous melanoma. Cochrane Database Syst Rev. 2023 Jan 17;1(1):CD012974. doi: 10.1002/14651858.CD012974.pub2. PMID 36648215

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three hundred forty-five participants were assessed for eligibility. Thirty-two participants were deemed ineligible for either not having measurable disease, per RECIST criteria (27 participants), or having an ineligible disease stage (5). The remaining 313 eligible participants were randomized.
Period: Step 1: Registration
Arm/Group | Arm I (Adjuvant Pembrolizumab) | Arm II (Adjuvant and Neoadjuvant Pembrolizumab)
Started | 159 | 154
Completed | 151 | 127
Not Completed | 8 | 27
Not completed — Still receiving protocol therapy | 0 | 10
Not completed — Withdrawal by Subject | 7 | 2
Not completed — Toxicity | 0 | 1
Not completed — Disease Progression | 0 | 12
Not completed — Co-morbidities | 0 | 1
Not completed — Scheduling Issues | 1 | 0
Not completed — Participant Refusal | 0 | 1
Period: Step 2: Surgery
Arm/Group | Arm I (Adjuvant Pembrolizumab) | Arm II (Adjuvant and Neoadjuvant Pembrolizumab)
Started | 151 | 127
Completed | 130 | 109
Not Completed | 21 | 18
Not completed — Participant Refusal | 2 | 1
Not completed — Neoadjuvant Toxicity | 0 | 3
Not completed — Metastatic Disease | 16 | 9
Not completed — Residual Disease | 2 | 1
Not completed — Trial Closed due to Covid-19 | 0 | 1
Not completed — Concerns about Exposure to Covid-19 | 0 | 1
Not completed — Disease other than melanoma identified at surgery | 0 | 2
Not completed — Radiotherapy-related Delays | 1 | 0
Period: Step 3: Adjuvant Pembrolizumab
Arm/Group | Arm I (Adjuvant Pembrolizumab) | Arm II (Adjuvant and Neoadjuvant Pembrolizumab)
Started | 130 | 109
Completed | 38 | 50
Not Completed | 92 | 59
Not completed — Still receiving protocol therapy | 41 | 33
Not completed — Disease Progression | 41 | 9
Not completed — Death | 4 | 1
Not completed — Other, unspecified reasons | 6 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Adjuvant Pembrolizumab) | Arm II (Adjuvant and Neoadjuvant Pembrolizumab) | Total
Number analyzed (Participants) | 159 | 154 | 313
Age, Continuous [Median (Full Range); unit: years] | 62 [22 to 88] | 64 [19 to 90] | 64 [19 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 62 | 110
  Male | 111 | 92 | 203
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 9 | 13
  Not Hispanic or Latino | 151 | 136 | 287
  Unknown or Not Reported | 4 | 9 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 150 | 141 | 291
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 4 | 10 | 14
Zubrod Performance Status Score [Count of Participants; unit: Participants] — Zubrod's performance-status scores range from 0 to 5, with higher scores indicating greater disability; a score of 0 indicates that the participant is fully active, 1 that the patient is restricted in strenuous activity but is ambulatory, and 2 that the participant is unable to work but is ambulatory and capable of self-care and up and about more than 50% of waking hours.
  Participants
    0 | 125 | 113 | 238
    1 | 33 | 39 | 72
    2 | 0 | 1 | 1
    Missing/Not Reported | 1 | 1 | 2
LDH Level [Count of Participants; unit: Participants] — LDH denotes lactate dehydrogenase.
  Participants
    Low or Normal | 138 | 132 | 270
    High | 21 | 22 | 43
Disease Stage [Count of Participants; unit: Participants] — Stages are defined according to the American Joint Committee on Cancer 'Cancer Staging Manual', 8th edition.
  Participants
    IIIB | 64 | 62 | 126
    IIIC | 74 | 69 | 143
    IIID | 10 | 9 | 19
    IV | 11 | 14 | 25
Primary Melanoma Subtype [Count of Participants; unit: Participants]
  Cutaneous or Unknown | 153 | 143 | 296
  Acral | 5 | 4 | 9
  Mucosal | 0 | 4 | 4
  Missing/Not Reported | 1 | 3 | 4
Ulceration [Count of Participants; unit: Participants]
  Yes | 46 | 56 | 102
  No | 58 | 50 | 108
  Unknown | 55 | 46 | 101
  Missing/Not Reported | 0 | 2 | 2
BRAF Mutation Status [Count of Participants; unit: Participants]
  Mutated | 38 | 41 | 79
  Wild-type | 64 | 62 | 126
  Unknown | 57 | 51 | 108
Previous BRAF and MEK Adjuvant Therapy [Count of Participants; unit: Participants]
  Yes | 1 | 3 | 4
  No | 158 | 151 | 309
Previous Radiotherapy [Count of Participants; unit: Participants]
  Yes | 1 | 2 | 3
  No | 158 | 152 | 310

OUTCOME MEASURES:

1. Primary Outcome: Two-Year Event-Free Survival Rate
Description: Event-free survival (EFS) is measured from date of randomization to date of first: documentation of progression that render participant unable to receive planned protocol surgery, off protocol therapy for any reason without subsequent protocol surgery, failure to begin adjuvant therapy within 84 days after surgery, relapse after surgery or death due to any cause. Participants last known to be alive and event-free are censored at date of last contact. All events that occurred before the start of adjuvant therapy were assigned an event date of 84 days.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Adjuvant Pembrolizumab) | Arm II (Adjuvant and Neoadjuvant Pembrolizumab)
Number analyzed (Participants) | 159 | 154
percentage of participants | 49 [41 to 59] | 72 [64 to 80]
Statistical Analysis 1: Comparison: Arm I (Adjuvant Pembrolizumab) vs Arm II (Adjuvant and Neoadjuvant Pembrolizumab); Test type: Superiority; p = 0.004, Log Rank; Hazard Ratio (HR) = 0.64

2. Secondary Outcome: Number of Participants With Grade 3 Through 5 Adverse Events That Are Related to Study Drug
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Duration of treatment and follow-up until relapse, death, or 3.5 years post randomization.
Population: Eligible participants that received protocol treatment
Measure: Number; unit: Participants
Groups:
- Arm I (Adjuvant Pembrolizumab): Within 17 days (preferably within 14 days) days after IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 18 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood throughout the study and MRI or CT on study.
  Biospecimen Collection: Undergo collection of blood Computed Tomography: Undergo CT Magnetic Resonance Imaging: Undergo MRI Pembrolizumab: Given IV Therapeutic Conventional Surgery: Undergo surgery
- Arm II (Adjuvant and Neoadjuvant Pembrolizumab): Patients receive pembrolizumab IV over 30 minutes on day 1 every 3 weeks for 3 cycles, then undergo surgery within 3 weeks. Within 84 days, patients receive pembrolizumab IV over 30 minutes every 3 weeks for 15 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood throughout the study and MRI or CT on study.
  Biospecimen Collection: Undergo collection of blood Computed Tomography: Undergo CT Magnetic Resonance Imaging: Undergo MRI Pembrolizumab: Given IV Therapeutic Conventional Surgery: Undergo surgery
Arm/Group | Arm I (Adjuvant Pembrolizumab) | Arm II (Adjuvant and Neoadjuvant Pembrolizumab)
Number analyzed (Participants) | 141 | 152
Participants
  Adrenal insufficiency | 0 | 1
  Alanine aminotransferase increased | 3 | 5
  Alkaline phosphatase increased | 0 | 1
  Anemia | 0 | 1
  Arthralgia | 1 | 0
  Arthritis | 1 | 0
  Aspartate aminotransferase increased | 2 | 4
  Blood and lymphatic system disorders - Other, spec | 1 | 0
  Cardiac disorders - Other, specify | 1 | 0
  Cardiac troponin I increased | 0 | 1
  Chest wall pain | 1 | 0
  Cognitive disturbance | 1 | 0
  Colitis | 0 | 1
  Dehydration | 0 | 1
  Diarrhea | 1 | 2
  Electrocardiogram QT corrected interval prolonged | 0 | 1
  Fall | 0 | 1
  Fatigue | 2 | 0
  Febrile neutropenia | 1 | 0
  Fever | 0 | 2
  Gallbladder infection | 1 | 0
  Headache | 0 | 1
  Hematoma | 1 | 0
  Hepatobiliary disorders - Other, specify | 1 | 0
  Hyperglycemia | 3 | 2
  Hypertension | 2 | 3
  Hypokalemia | 0 | 2
  Hyponatremia | 0 | 1
  Hypothyroidism | 1 | 0
  Infections and infestations - Other, specify | 1 | 0
  Lung infection | 0 | 2
  Lymphocyte count decreased | 3 | 0
  Metabolism and nutrition disorders - Other, specif | 1 | 0
  Myalgia | 1 | 0
  Myocarditis | 1 | 2
  Myositis | 1 | 0
  Nausea | 0 | 2
  Neutrophil count decreased | 0 | 1
  Platelet count decreased | 1 | 0
  Pneumonitis | 0 | 2
  Pruritus | 2 | 1
  Rash maculo-papular | 4 | 2
  Respiratory failure | 1 | 0
  Sepsis | 0 | 1
  Seroma | 1 | 1
  Skin and subcutaneous tissue disorders - Other, sp | 0 | 1
  Skin infection | 1 | 1
  Small intestinal obstruction | 1 | 0
  Soft tissue infection | 0 | 1
  Stroke | 0 | 1
  Surgical and medical procedures - Other, specify | 0 | 1
  Syncope | 1 | 2
  Thromboembolic event | 1 | 1
  Urinary tract infection | 1 | 1
  Vomiting | 0 | 1
  White blood cell decreased | 0 | 1
  Wound dehiscence | 0 | 1
  Wound infection | 0 | 2

3. Secondary Outcome: Two-Year Overall Survival Rate
Description: Overall survival (OS) is measured from date of randomization to date of death due to any cause. Participants known to be alive are censored at date of last contact.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Adjuvant Pembrolizumab) | Arm II (Adjuvant and Neoadjuvant Pembrolizumab)
Number analyzed (Participants) | 159 | 154
percentage of participants | 79 [71 to 89] | 87 [80 to 95]

4. Secondary Outcome: Response Rate
Description: On the neoadjuvant arm, the response rate was assessed after neoadjuvant therapy and before surgical resection. The response rate includes both complete response (CR) and partial response (PR). CR is defined as complete disappearance of all target and non-target lesions, no new lesions, and no disease related symptoms. PR is defined as greater than or equal to 30% decrease under baseline of the sum of all appropriate diameters of all target measurable lesions, no unequivocal progression or non-measurable disease, and no new lesions. The best response rate is calculated from the sequence of objective statuses. CR is defined as two or more objective statuses of CR a minimum of four weeks apart documented before progression or symptomatic deterioration. PR is defined as two or more objective statuses of PR or better a minimum of four weeks apart documented before progression or symptomatic deterioration, but not qualifying as CR.
Time Frame: 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Number of Participants Receiving Surgery
Description: To determine the number of participants on each arm who received the surgery planned at randomization.
Time Frame: 2.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Adjuvant Pembrolizumab) | Arm II (Adjuvant and Neoadjuvant Pembrolizumab)
Number analyzed (Participants) | 159 | 154
Participants | 151 | 127

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow-up until relapse, death, or 3.5 years post randomization
Description: AEs and SAEs are reported by CTCAE v5.0. 152 participants on the neoadjuvant arm and 141 participants on the adjuvant arm that were eligible and received some protocol treatment were evaluable for AEs. 154 eligible participants on the neoadjuvant arm and 159 eligible participants on the adjuvant arm were analyzed for all-cause mortality.
Arm/Group | Arm I (Adjuvant Pembrolizumab) | Arm II (Adjuvant and Neoadjuvant Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 22/159 | 14/154
Serious Adverse Events (participants affected / at risk) | 33/141 | 34/152
Other Adverse Events (participants affected / at risk) | 132/141 | 148/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Adjuvant Pembrolizumab) (N=141) | Arm II (Adjuvant and Neoadjuvant Pembrolizumab) (N=152)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Cardiac disorders-Other (Cardiac disorders) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 2
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Endocrine disorders-Other (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 0 | 3
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3
Edema limbs (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 0
Fever (General disorders) | 1 | 8
Flu like symptoms (General disorders) | 1 | 0
General disorders and administration site conditio (General disorders) | 0 | 1
Hypothermia (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatobiliary disorders-Other (Hepatobiliary disorders) | 1 | 0
Gallbladder infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 3
Sepsis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 3 | 2
Soft tissue infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Injury, poisoning and procedural complications-Oth (Injury, poisoning and procedural complications) | 0 | 2
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 4
Alkaline phosphatase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 5
Creatinine increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Metabolism and nutrition disorders-Other (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasms benign, malignant and unspecified (incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0
Facial muscle weakness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 2
Stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Transient ischemic attacks (Nervous system disorders) | 1 | 0
Vasovagal reaction (Nervous system disorders) | 1 | 1
Pregnancy, puerperium and perinatal conditions-Oth (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Personality change (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Hematoma (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 1
Lymph leakage (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Adjuvant Pembrolizumab) (N=141) | Arm II (Adjuvant and Neoadjuvant Pembrolizumab) (N=152)
Anemia (Blood and lymphatic system disorders) | 37 | 54
Blood and lymphatic system disorders-Other (Blood and lymphatic system disorders) | 8 | 10
Eosinophilia (Blood and lymphatic system disorders) | 10 | 6
Hyperthyroidism (Endocrine disorders) | 11 | 6
Hypothyroidism (Endocrine disorders) | 26 | 26
Blurred vision (Eye disorders) | 6 | 10
Eye disorders-Other (Eye disorders) | 7 | 10
Abdominal pain (Gastrointestinal disorders) | 9 | 14
Constipation (Gastrointestinal disorders) | 19 | 22
Diarrhea (Gastrointestinal disorders) | 34 | 39
Dry mouth (Gastrointestinal disorders) | 15 | 7
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 6 | 11
Nausea (Gastrointestinal disorders) | 33 | 40
Vomiting (Gastrointestinal disorders) | 13 | 18
Chills (General disorders) | 13 | 11
Edema limbs (General disorders) | 33 | 39
Fatigue (General disorders) | 90 | 90
Fever (General disorders) | 10 | 10
Pain (General disorders) | 33 | 33
Infections and infestations-Other (Infections and infestations) | 17 | 13
Skin infection (Infections and infestations) | 15 | 15
Upper respiratory infection (Infections and infestations) | 3 | 8
Urinary tract infection (Infections and infestations) | 8 | 5
Seroma (Injury, poisoning and procedural complications) | 11 | 7
Alanine aminotransferase increased (Investigations) | 17 | 27
Alkaline phosphatase increased (Investigations) | 13 | 21
Aspartate aminotransferase increased (Investigations) | 17 | 29
Blood bilirubin increased (Investigations) | 8 | 13
Creatinine increased (Investigations) | 17 | 28
Investigations-Other (Investigations) | 8 | 5
Lymphocyte count decreased (Investigations) | 19 | 30
Platelet count decreased (Investigations) | 9 | 13
Thyroid stimulating hormone increased (Investigations) | 10 | 16
Weight loss (Investigations) | 18 | 13
White blood cell decreased (Investigations) | 8 | 11
Anorexia (Metabolism and nutrition disorders) | 15 | 27
Hypercalcemia (Metabolism and nutrition disorders) | 8 | 9
Hyperglycemia (Metabolism and nutrition disorders) | 46 | 48
Hyperkalemia (Metabolism and nutrition disorders) | 6 | 13
Hypoalbuminemia (Metabolism and nutrition disorders) | 12 | 19
Hypocalcemia (Metabolism and nutrition disorders) | 18 | 9
Hypoglycemia (Metabolism and nutrition disorders) | 6 | 8
Hypokalemia (Metabolism and nutrition disorders) | 9 | 18
Hyponatremia (Metabolism and nutrition disorders) | 23 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 | 29
Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 19 | 17
Neck pain (Musculoskeletal and connective tissue disorders) | 10 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 | 29
Dizziness (Nervous system disorders) | 13 | 14
Dysgeusia (Nervous system disorders) | 8 | 6
Headache (Nervous system disorders) | 23 | 29
Paresthesia (Nervous system disorders) | 20 | 18
Peripheral sensory neuropathy (Nervous system disorders) | 9 | 9
Anxiety (Psychiatric disorders) | 8 | 16
Insomnia (Psychiatric disorders) | 13 | 13
Urinary frequency (Renal and urinary disorders) | 8 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 30
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 23 | 20
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Dry skin (Skin and subcutaneous tissue disorders) | 14 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 36 | 43
Rash acneiform (Skin and subcutaneous tissue disorders) | 9 | 10
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 42 | 44
Skin and subcutaneous tissue disorders-Other (Skin and subcutaneous tissue disorders) | 26 | 25
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 8 | 12
Surgical and medical procedures-Other (Surgical and medical procedures) | 2 | 8
Hypertension (Vascular disorders) | 40 | 44
Lymphedema (Vascular disorders) | 15 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT03698019/Prot_SAP_000.pdf